CLINICAL TRIAL: NCT07382180
Title: More Than Weight Loss: Real-World Tirzepatide Use in Post-Bariatric Weight Regain and Preoperative Obesity Care
Brief Title: Real-World Tirzepatide Therapy in Post-Bariatric Weight Regain and Preoperative Obesity Patients
Acronym: TIR-REAL
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, surgeon, Azienda Sanitaria Locale Napoli 2 Nord
Other Study IDs: 11182022
Record Dates: First submitted 2026-01-26; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight; Weight Regain; Obesity, Morbid
Keywords: Obesity; Weight Regain; Obesity, Morbid
MeSH Terms: conditions — Obesity; Overweight; Obesity, Morbid | interventions — Obesity Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Post-Bariatric Weight Regain: Adult patients with a history of sleeve gastrectomy who developed clinically significant weight regain, defined as an increase of at least 25% from the postoperative nadir weight, and who were treated with tirzepatide as part of routine clinical care.
  Interventions: Drug: Tirzepatide is administered as part of routine clinical care for obesity management, according to standard prescribing practices. Dosing and treatment duration are determined by the treating physician
- Preoperative Obesity Management: Adult patients with obesity receiving tirzepatide as part of preoperative medical optimization before planned bariatric or metabolic surgery, managed according to standard clinical practice.
  Interventions: Drug: Tirzepatide is administered as part of routine clinical care for obesity management, according to standard prescribing practices. Dosing and treatment duration are determined by the treating physician

INTERVENTIONS:
Drug: Tirzepatide is administered as part of routine clinical care for obesity management, according to standard prescribing practices. Dosing and treatment duration are determined by the treating physician — This study is conducted as a non-interventional, investigator-initiated observational study using data collected during routine clinical practice. No randomization, blinding, or protocol-mandated procedures are applied. Treatment decisions, follow-up schedules, and clinical assessments are determined solely by the treating physicians according to standard care. Data are collected retrospectively and prospectively from clinical records and routine follow-up visits. The study does not alter patient management and does not involve additional risks beyond usual clinical practice.

SUMMARY:
This multicenter retrospective observational study evaluates the real-world use of tirzepatide in adult patients with post-bariatric weight regain and in patients with obesity undergoing preoperative management. The study analyzes changes in body weight and metabolic parameters, as well as treatment tolerability and safety, during routine clinical care. No experimental interventions are performed, and all patients receive tirzepatide as part of standard medical practice.

DETAILED DESCRIPTION:
Obesity is a chronic and progressive disease that often requires long-term management. Although bariatric surgery is an effective treatment for severe obesity, a significant proportion of patients experience weight regain several years after surgery. In addition, many patients with obesity require medical treatment before surgery to reduce surgical risk and improve perioperative outcomes. In both situations, there is a growing need for effective and well-tolerated pharmacological therapies that can be integrated into routine clinical care.

Tirzepatide is a dual glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide-1 (GLP-1) receptor agonist that has demonstrated significant effects on body weight reduction and metabolic control. While its efficacy has been established in randomized clinical trials, data on its use in real-world clinical practice, particularly in post-bariatric patients with weight regain and in patients undergoing preoperative obesity management, are still limited.

This multicenter observational cohort study evaluates the real-world use of tirzepatide in adult patients managed within routine bariatric and metabolic care pathways. The study includes two patient populations: individuals with clinically significant weight regain after sleeve gastrectomy and patients with obesity treated with tirzepatide as part of preoperative medical optimization before planned surgical intervention. All patients receive tirzepatide according to standard clinical practice, without any experimental procedures or protocol-mandated treatment changes.

Clinical, anthropometric, and metabolic data are collected at baseline and during scheduled follow-up visits, in accordance with routine care. The primary objective is to assess changes in body weight over time. Secondary objectives include evaluation of metabolic parameters, treatment tolerability, and the occurrence of adverse events. Safety data are collected as part of standard clinical monitoring.

By analyzing outcomes in a real-world setting, this study aims to provide clinically meaningful evidence on the effectiveness and safety of tirzepatide outside of controlled trial environments. The results are intended to support clinicians in decision-making for the management of obesity in complex clinical scenarios, such as post-bariatric weight regain and preoperative optimization, and to better define the role of pharmacological therapy as part of an integrated, long-term obesity care strategy.

ELIGIBILITY:
nclusion Criteria

* Adult patients aged 18 years or older.
* Diagnosis of obesity, defined according to standard clinical criteria, managed within a bariatric and metabolic care pathway.
* Initiation of tirzepatide therapy at a starting dose of 5 mg as part of routine clinical practice.
* Allocation to one of the following clinical cohorts:
* Patients with prior sleeve gastrectomy and clinically significant weight regain, defined as a ≥25% increase in body weight relative to the postoperative nadir weight, with a minimum interval of 36 months from surgery; or
* Patients with obesity undergoing preoperative medical optimization prior to planned bariatric surgery.
* Availability of complete baseline clinical and anthropometric data at treatment initiation.
* Planned clinical follow-up for at least 6 months after initiation of tirzepatide therapy.
* Ability to provide written informed consent for the use of clinical data for research purposes, according to local regulations.

Exclusion Criteria

* Age younger than 18 years.
* Prior bariatric procedures other than sleeve gastrectomy (for the weight regain cohort).
* Current or previous treatment with tirzepatide before study enrollment.
* Use of other anti-obesity pharmacological agents during the observation period.
* Contraindications to tirzepatide therapy according to the approved product label.
* Pregnancy or breastfeeding at the time of treatment initiation or during follow-up.
* Presence of severe medical, psychiatric, or cognitive conditions that, in the investigator's judgment, could interfere with adherence to treatment or follow-up assessments.
* Incomplete baseline data or anticipated inability to complete the planned 6-month follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients with obesity managed within established bariatric and metabolic care pathways at participating referral centers. Participants are selected from individuals who initiate tirzepatide therapy as part of routine clinical practice, either for medical optimization prior to planned bariatric surgery or for the management of clinically significant weight regain following prior sleeve gastrectomy.
  All participants receive standard multidisciplinary care, including medical, nutritional, and metabolic evaluation, and are followed longitudinally through scheduled outpatient visits. The study population reflects a real-world clinical setting and includes patients with a broad range of obesity-related metabolic profiles, representative of routine bariatric practice.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01-18 (Actual); Study Completion 2026-01-18 (Actual)

PRIMARY OUTCOMES:
Percentage Total Body Weight Loss (%TBWL) | From baseline (initiation of tirzepatide therapy) to 6 months of treatment
  Percentage total body weight loss (%TBWL) was calculated as the percentage change in body weight from baseline to 6 months after initiation of tirzepatide therapy. Baseline body weight was defined as the body weight recorded at the start of treatment. Body weight measurements were obtained during scheduled outpatient visits using calibrated clinic scales, with participants wearing light clothing and no shoes.
  %TBWL was calculated using the following formula: [(baseline body weight - follow-up body weight) / baseline body weight] × 100.
  This outcome measure was selected as a standardized and clinically meaningful indicator of treatment effectiveness in obesity management, allowing comparison of weight reduction across patients with different baseline body weights and clinical indications.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | From baseline (initiation of tirzepatide therapy) to 6 months of treatment
  Change in body mass index (BMI) from baseline to 6 months after initiation of tirzepatide therapy. BMI was calculated as body weight in kilograms divided by height in meters squared (kg/m²). Baseline BMI was defined as the value recorded at treatment initiation. Body weight and height were measured during outpatient visits using calibrated clinical equipment.
Safety and Tolerability of Tirzepatide | From baseline (initiation of tirzepatide therapy) to 6 months of treatment
  Incidence and type of treatment-emergent adverse events during tirzepatide therapy, including gastrointestinal symptoms and treatment discontinuation due to adverse effects. Adverse events were collected through clinical visits and review of medical records and were classified according to routine clinical practice.
Change in Mood Status | From baseline (initiation of tirzepatide therapy) to 6 months of treatment
  Change from baseline to 6 months in self-reported mood status, assessed during routine outpatient visits using the Patient Global Mood Assessment (PGMA), a standardized, non-diagnostic patient-reported outcome measure evaluating overall mood and emotional well-being.
  The Patient Global Mood Assessment (PGMA) is scored on a 7-point Likert scale, ranging from -3 (marked worsening of mood) to +3 (marked improvement of mood), with 0 indicating no change compared with baseline.
  Higher scores indicate improvement in mood and emotional well-being, while lower scores indicate worsening.

CONTACTS AND LOCATIONS:
Locations (1):
- Head of bariatric surgery, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No
This is an observational real-world study based on data collected during routine clinical care. Individual participant data are derived from medical records and are subject to data protection and privacy regulations. No formal plan for sharing individual participant data has been established, as data analyses are conducted on de-identified, aggregated datasets to ensure confidentiality and regulatory compliance.